CLINICAL TRIAL: NCT07296107
Title: Leveraging IVF to Identify Prenatal Effects Independent of Shared Maternal-Child Genes
Brief Title: In Vitro Fertilization (IVF) and Prenatal Effects Independent of Genetics
Status: Not yet recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: University of California, Los Angeles (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Catherine Monk, Diana Vagelos Professor of Women's Mental Health, Columbia University
Other Study IDs: AAAV4123; 1R01HD118949-01 (NIH)
Record Dates: First submitted 2025-12-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Maternal Distress; Child Development
Keywords: Developmental Origins of Health and Disease (DOHaD); Maternal Health; Child development; IVF
MeSH Terms: conditions — Developmental Origins of Health and Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cord blood, placenta, maternal blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Donor Oocyte/Embryo IVF Pregnancies: This cohort includes pregnant individuals who conceived through in vitro fertilization (IVF) using donor oocytes or embryos, and are therefore not genetically related to the fetus. Participants follow the same study protocol as the non donor oocyte cohort, with enrollment in the second trimester and data collection through delivery and early postpartum. The purpose of including this cohort is to evaluate the effects of maternal prenatal distress and well-being on perinatal development independent of shared maternal-child genetics. Data collection includes psychosocial questionnaires, maternal physiological monitoring, blood draws for immune and transcriptomic analyses, placental and cord blood collection at delivery, newborn physiological monitoring during the postpartum hospital stay, and birth outcomes obtained from the electronic health record (EHR).
  Interventions: Other: Prenatal maternal psychosocial and biological assessment protocol
- Non-Donor Oocyte IVF Pregnancies: This cohort includes pregnant individuals who conceived through IVF using their own oocytes, and are therefore genetically related to the fetus. Participants follow the same study protocol as the donor oocyte cohort, with enrollment in the second trimester and data collection through delivery and early postpartum. This group serves as a comparison to assess whether observed associations between maternal prenatal distress, biological markers, and infant neurodevelopment are attributable to intrauterine (environmental) influences or shared genetic factors. Data collection includes psychosocial questionnaires, maternal physiological monitoring, blood draws for immune and transcriptomic analyses, placental and cord blood collection at delivery, newborn physiological monitoring during the postpartum hospital stay, and birth outcomes obtained from the electronic health record (EHR)
  Interventions: Other: Prenatal maternal psychosocial and biological assessment protocol

INTERVENTIONS:
Other: Prenatal maternal psychosocial and biological assessment protocol — This is not a therapeutic or experimental intervention. The data-collection protocol includes structured psychosocial questionnaires, physiological monitoring, maternal blood draws, placental and cord blood collection, and newborn physiological monitoring. These procedures are used to observe associations between maternal prenatal distress and infant outcomes. All participants undergo the same assessments; no clinical treatment or behavioral manipulation is delivered.

SUMMARY:
This study examines how maternal stress during pregnancy affects infant brain and behavioral development, focusing on whether these effects are due to the prenatal environment or shared genes. By comparing IVF pregnancies using donor eggs/embryos (no shared genetics) with non-donor IVF pregnancies, the investigators aim to understand how stress influences the baby's development independent of genetic factors.

Participants will complete questionnaires, provide blood samples, and take part in placenta and cord blood collection, fetal monitoring, and newborn brain activity assessments.

Aim 1: The influence of maternal distress on perinatal neurobehavioral development.

Hypotheses: Independent of IVF group status, higher maternal AL will be associated with higher 3rd trimester FHR reactivity, lower FHR variability, AND lower FHR-movement coupling

Aim 2: Maternal distress affecting placenta gene methylation.

Hypotheses: Independent of IVF group status, maternal AL will be associated with placenta differential DNA methylation in glucocorticoid-regulating genes (FKBP5 and HSD11B2),

Aim 3: Maternal experiences associated with unique placenta transcriptomic profiles.

Hypotheses: Independent of IVF group status, maternal AL and well-being each will be associated with unique placenta gene expression in pro-inflammatory genes

DETAILED DESCRIPTION:
To rigorously test the Developmental Origins of Health and Disease (DOHaD) research model, this project will leverage the spectacular scientific advancements of in vitro fertilization (IVF) and compare maternal prenatal distress effects between IVF donor oocyte/embryo and non-donor oocyte pregnancies. This will be the first study to use multidisciplinary (neurobehavioral, epigenetic, transcriptomic) methods with adoption-at-conception pregnant individuals to determine whether prenatal programming can be detected independent of shared maternal-child genes.

Decades of prospective DOHaD research with birthing individuals and their genetic children, including reports from our group, support the prenatal programming hypothesis that pregnant individuals' mental health affects the next generation's. Seminal, population-based studies using parent reports, such as the Avon Longitudinal Study of Parents and Children (ALSPAC), showed pregnant women in the top 15% for anxiety symptoms had children with nearly twice the risk of mental health disorders across ages 4-13 after controlling for confounders including postpartum depression. In our work and others' using objective assessments, maternal prenatal distress associated with higher 3rd trimester fetal heart rate (FHR) reactivity, from EEG in newborns lower high- frequency power and greater frontal asymmetry (itself associated with adult depression), and decrements in NIH ToolBox executive functioning and motor skills at 4-8 years old. However, for each of these findings, shared maternal-child genes cannot be ruled out. Animal models - in which the genetic background and stress exposure can be manipulated - show prenatal stress leads to anxious and depressed behavioral phenotypes independent of genetic inheritance, though limitations in the applicability to humans include: stressors' ecological validity, differences in gestational biology, and developmental timing. Genetically-informed studies, including those with donor IVF participants, show mixed evidence for prenatal distress effects. However, designs are frequently retrospective, including in IVF research, such that medical confounds also are not well controlled. Mechanistic approaches, such as our work and others' work focused on the placenta, a gestational organ at the maternal-fetal interface, show maternal distress associated with epigenetic regulation of placenta glucocorticoid and pro-inflammatory genes and child outcomes; to date, no study using IVF to circumvent genetic confounding has included mechanistic approaches. Finally, most DOHaD science concerns maternal distress effects; to advance prenatal programming research and enhance its relevance for clinical interventions, maternal social connection and other aspects of well-being also should be examined. Our study will address these design limitations and aim to identify maternal prenatal distress effects independent of shared maternal-child genes.

In a longitudinal study of 2nd trimester pregnant individuals (60 donor oocyte/embryo,120 non-donor oocyte), n=180 post attrition, protocol is: Zoom-based psychosocial questionnaires 26-28 weeks (Pregnancy Session 1); laboratory session for maternal EKG, blood pressure, blood draw (immune markers), psychosocial questionnaires, fetal neurobehavior 34-36 weeks (Pregnancy Session 2); collect placenta and cord blood (cortisol); newborn EEG in hospital; medical record data; and, methods: placenta targeted/genome-wide methylation, gene expression, distress, Allostatic Load (AL): Test three aims, identifying, independent of IVF group status.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals at 22-26 gestational weeks with donor and homologous IVF pregnancies, ages 18-50.
2. Participants must be patients receiving their perinatal health care through Columbia University Irving Medical Center's Department of OB/GYN and delivering at New York-Presbyterian Morgan Stanley Children's Hospital.
3. Participants will include the offspring of patients receiving care at the above institutions.
4. Enrollment Location(s): Columbia University Irving Medical Center's Department of OB/GYN, delivering at New York-Presbyterian Morgan Stanley Children's Hospital.

Exclusion Criteria:

1. Current cigarette smoking
2. Active drug use
3. Unstable psychiatric condition
4. Multiple fetal pregnancy
5. Known chromosomal, genetic, or major fetal malformations (unlikely due to routine preimplantation genetic testing)
6. Inflammatory conditions including rheumatoid arthritis, lupus, and multiple sclerosis
7. Current use of synthetic glucocorticoids
8. Not planning to deliver at a CUIMC-affiliated hospital

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This five-year study will recruit and enroll approximately 200 pregnant individuals, ages 18-50 years, using IVF (120 homologous, 60 donor oocyte/embryo) and their offspring to achieve a post-attrition sample size of n=180. While based in Washington Heights, the sample reflects individuals undergoing IVF, not the general neighborhood. Based on Columbia Fertility Center data and national IVF trends, the investigators expect participants to be mostly Non-Hispanic/Latinx. While the investigators aim for inclusivity and diversity, non-English speakers will not be enrolled due to study team language constraints.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in fetal heart rate (FHR) | At Pregnancy Session 2 (approximately 34-36 weeks of pregnancy)
  This is to measure 3rd trimester fetal heart rate (FHR) reactivity. Change in FHR in response to maternal response to the Stroop task, indicating greater fetal autonomic response associated with maternal distress. Units: Beats per minute (bpm). Greater FHR indicates higher stress.
Standard deviation of fetal heart rate | At Pregnancy Session 2 (approximately 34-36 weeks of pregnancy)
  This is to measure fetal heart rate (FHR) variability, reflecting less vagal modulation of the heart associated with maternal distress. Units: Standard deviation of beats per minute. Lesser standard deviation (SD) indicates lower stress.
Cross correlation of fetal movement and heart rate change | At Pregnancy Session 2 (approximately 34-36 weeks of pregnancy)
  This is to measure fetal heart rate (FHR)-movement coupling, reflecting central nervous system regulation. Units: Cross correlation value. Lower value indicates lower coupling.
Average percent DNA methylation of the FKBP5 gene in placental tissue | At delivery (approximately 37-40 weeks)
  This is to measure FKBP5 DNA Methylation. Units: proportion of methylated vs unmethylated. Greater percent indicates higher methylation.
Average percent DNA methylation of the HSD11B2 gene in placental tissue | At delivery (approximately 37-40 weeks)
  This is to measure HSD11B2 DNA Methylation. Units: proportion of methylated vs unmethylated. Greater percent indicates higher methylation.
Relative expression of key pro-inflammatory markers in placental tissue | At delivery (approximately 37-40 weeks)
  This is to measure expression of Pro-Inflammatory Placental Genes. Units: Gene expression. Greater value indicates greater expression.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Monk, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided